CLINICAL TRIAL: NCT01425411
Title: Effect of Valsartan on Left Ventricular Myocardial Functions in Hypertensive Patients With Left Ventricular Hypertrophy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Nagehan Kucukler, MD, Mustafa Kemal University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: vals262626
Record Dates: First submitted 2011-08-18; First posted 2011-08-30 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Hypertension; Left Ventricular Hypertrophy
Keywords: hypertension; left ventricular hypertrophy; angiotensin receptor blocker; midwall mechanics; tissue Doppler imaging; Hypertension with left ventricular hypertrophy
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular | interventions — Valsartan

ARMS (1):
- Valsartan treatment (Experimental)
  Interventions: Drug: valsartan

INTERVENTIONS:
Drug: valsartan — 80/160 mg dosage of valsartan or 160+12,5 mg valsartan+hydrochlorothiazide combination, once a day, for six months
  Other Names: Diovan 80 mg; Diovan 160 mg; Co-diovan 160/12,5 mg

SUMMARY:
The study hypothesis: Valsartan as an angiotensin II receptor blocker treatment has beneficial effects on both midwall mechanics and myocardial functions in hypertensive patients with Left ventricular hypertrophy.

ELIGIBILITY:
Inclusion Criteria:

* hypertension with left ventricular hypertrophy

Exclusion Criteria:

* clinical or laboratory evidence of secondary hypertension
* heart failure
* ischemic heart disease
* valvular heart disease
* arrhythmias
* peripheral vascular disease
* chronic obstructive pulmonary disease
* neurologic disorders
* diabetes mellitus
* renal dysfunction
* notable systemic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
change from baseline in midwall fractional shortening (mFS) and tissue Doppler systolic wave (Sm) measured by echocardiography at six months | six months

SECONDARY OUTCOMES:
change from baseline in systolic and diastolic blood pressure at six months | six months
change from baseline in left ventricular mass index measured by echocardiography at six months | six months

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Yalcin, M.D., Principal Investigator — Mustafa Kemal University: Turkey
Locations (1):
- Mustafa Kemal University School of Medicine, Department of Cardiology, Antioch, Antioch, Turkey (Türkiye)

REFERENCES:
- [Derived] Kucukler N, Kurt IH, Topaloglu C, Gurbuz S, Yalcin F. The effect of valsartan on left ventricular myocardial functions in hypertensive patients with left ventricular hypertrophy. J Cardiovasc Med (Hagerstown). 2012 Mar;13(3):181-6. doi: 10.2459/JCM.0b013e3283511f00. PMID 22306782